CLINICAL TRIAL: NCT05564559
Title: Multifamily Group Psychoeducation for Substance Use Disorders: A Non-randomized Controlled Trial in Turkey
Brief Title: Multifamily Group Psychoeducation for SUD's in Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, BEYZA NUR KAYTAZ YILMAZ, Principal Investigator, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE-BNKY-001
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Disease; Mental Disorders, Severe; Substance-Related Disorders; Substance Use Disorders; Alcohol Use Disorder
Keywords: multi-family psychoeducation; substance abuse disorder; group psychoeducation; group study; family psychoeducation
MeSH Terms: conditions — Disease; Mental Disorders; Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: It is a 2-arm, non-randomized clinical study consisting of an intervention and a control group (waiting list) aiming to provide 8 weeks of multi-family psychoeducation to the families of people living with a diagnosis of substance abuse disorder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFGP intervention (Experimental): This group will provide 8 weeks of multi-family psychoeducation to the families of people living with a diagnosis of substance abuse disorder.
  Interventions: Other: multifamily group psychoeducation
- Wait list-control group (No Intervention): This group will provide 8 weeks of multi-family psychoeducation to the families of people living with a diagnosis of substance abuse disorder after the intervention group is completed. This group is the control group on the waiting list.

INTERVENTIONS:
Other: multifamily group psychoeducation — The intervention involves 8 weeks of multifamily psychoeducation for families. Duration of sessions: 75 minutes on average Context: First session: psychoeducation on substance-abuse disorders; second session; effects of addiction on the family; third session; illness management; fourth session; supporting recovery; fifth session; improving stress coping skills/stress management; sixth session; developing problem-solving skills; seventh session; strengthening the family; eighth session; working with stigma Preferred approach: face-to-face, multi-family Approach: Psychoeducation
  Arms: MFGP intervention

SUMMARY:
The aim of this study is to investigate the effects of multi-family group psychoeducation (MFGP) on the families of people living with a diagnosis of substance abuse disorder on patients and their families.

It has been reported that families are affected by substance-related disorders. Families that are the target of psychoeducational practices for families are defined as follows: "Family" is a relative, biological family member, partner, close friend, or any other support person or a person who sees herself/himself as the patient's family. In most studies, it has been stated that including family members in the patient's treatment provides additional benefits to substance use services and makes long-term recovery more likely. Studies have found that MFGP is associated with fewer relapses and hospitalizations, improved family well-being, increased participation in vocational rehabilitation, higher employment rates, and reduced costs of care. Multifamily psychoeducation aims to increase the family's knowledge about substance use disorders and to include them in the recovery process.

Study Design:The intervention involves 8-week MFGP for families. During the 8 sessions, it was planned to conduct face-to-face psychoeducational group work, with each session lasting 75 minutes on average. The MFGP to be covered during 8 sessions was created by evaluating MFGP modules from 3 different sources.

Intervention protocols included these subjects:

First session: Psychoeducation on Substance-Abuse Disorders Second session: Effects of Addiction on the Family Third session: illness management Fourth session: Supporting Recovery Fifth session: Improving Stress Coping Skills/Stress Management Sixth session: Developing Problem-Solving Skills Seventh session: Strengthening the Family Eighth session: Working with Stigma

Study population: Families of people suffering from substance abuse disorders were studied.

Expected outcomes: An increase in general and social functionality, a decrease in depression, anxiety, and self-stigma, an increase in quality of life, and treatment compliance are expected for patients. For families, it is expected that depression, anxiety, self-stigma, and caregiving burnout decrease, funcitonalty and quality of life increases and people gain skills to cope with stress.

DETAILED DESCRIPTION:
Research Method:

The population of the research is all individuals who live in Istanbul and have a relative living with the diagnosis of substance-related disorder. The sample of the study is the families of people living with the diagnosis of substance use disorders. These families are receiving service from Maltepe University Faculty of Medicine AMATEM clinic in Istanbul.

The literature was reviewed to determine the effect size and sample size of the study. Considering the purpose, design, and target audience of the research, the study by Fiorillo et al. was accepted as a reference publication (Fiorillo et al. 2015). Based on the aforementioned study, the t test family calculated the difference between two dependent means (Matched Pair Test) f: 0.31 (exact value: 0.3144855) and the total number of samples was determined as 64. When loss rates are included, the reference publication Fiorillo et al. (2015) stated that the sample loss rate (attrition rate) was 7% for the intervention group and 6% for the control group. The participant loss rate was accepted as 10%. In this case, considering the power analysis and the loss rates in the reference publication, the final sample number for this study was determined as 70 in total, and 35 participants will form the intervention group and 35 participants will form the control group. 35 patient families and patients will be in the intervention group, and 35 patient families and patients will be in the control group. Patients will not receive any intervention, only data collection tools will be measured.

The sample will be selected from the population using the "Convenience Sampling Method'.Families will be informed about this study with the brochure that will be given to them during their outpatient clinic visits. Families who agree to participate in the study will first be presented with the 2 dates specified for the study's intervention and control group/waiting list. Whatever date is found suitable for the families, they will participate in the intervention or control group accordingly. The first set schedule will be the intervention group, and the second will be the control group/waiting list. No measurements will be made after the intervention to the waiting list/control group. During this period, all patients will receive standard treatment.

In the descriptive analysis of the data, the number, percentage, minimum, maximum, mean, and standard deviation values will be given. The Statistical Package for the Social Sciences (SPSS) 24.0 program will be used in the analysis of the data. The significance level will be set at p<0.05. An Analysis of Variance (ANOVA) test will be performed for repeated measurements.

Pre-Intervention: Introducing the study to families and giving informed consent forms to families are among the procedures at this stage. In addition, at this stage, a 45-minute pre-interview will be held in order to assign one of the intervention or control (waiting list) groups according to the working schedule of the families who agreed to participate in the study and to take pre-test measurements before the intervention.

Intervention: A previously standardized 8-week multi-family group psychoeducation protocol is applied to the intervention group. Meanwhile, the control group is on the waiting list.

Post-intervention: At the end of the intervention, post-tests are applied to the intervention group and control group. After this stage of the study, an intervention is also applied to the control group on the waiting list. The data collection phase of the study will be over after the intervention has been given to the intervention group and the post-test measurements have been made. No measurements will be taken after the intervention is applied to the control group.

ELIGIBILITY:
Inclusion Criteria

for patients:

* From 18 to 64 years old.
* Living with a diagnosis of substance use disorders according to DSM-5.
* Agree to be participants in the study.

for families:

-Identifying as a relative/family member of someone living with a substance use disorder.

Exclusion Criteria

for patients:

* Patients with impaired thinking and perception.
* Be over 65 years old. Having problems with Turkish language skills.
* Living with another physical illness that caused disability.
* Living with another severe mental illness that causes disability (Schizophrenia, schizoaffective disorder, epilepsy, etc.).

for families:

* Living with a mental disability.
* Living with a substance use disorder diagnosis.
* Having difficulties with Turkish language skills.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Families' Burden | The change scores of the control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  People with relatives living with serious mental illness may experience burnout due to caregiving. Eight weeks of multifamily psychoeducation is expected to reduce the burnout caused by caregiving. Caregiver burnout will be measured with the Zarit Caregiver Burden Scale. The scale, on which the burden of caregivers of individuals with serious mental illness is evaluated, consists of 19 items. The scale is in a 5-point Likert type and the score that can be obtained from the scale varies between 19 and 95 points. As the scores obtained from the scale increase, the severity of the burden also increases.

SECONDARY OUTCOMES:
Social Functioning | The change scores of the control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  Whether there is a change in the social functionality of the patients after 8 weeks of multifamily psychoeducation will be evaluated with the Social Functioning Assessment Scale. The scale, which evaluates social functionality in individuals with serious mental illness, consists of 19 items. The scale is in a 3-point Likert type and the score that can be obtained from the scale varies between 19 and 57. A high score on the scale means that the person's functionality is high.

OTHER OUTCOMES:
Quality of Life Assessment | The change scores of the families' control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  At the end of multi-family psychoeducation, the change in the quality of life of families will be measured. Changes in health-related quality of life will be assessed with WHOQOL-BREF-TR. The scale measuring the quality of life in individuals consists of 27 items. The scale is in a 5-point Likert type and the score that can be obtained from the scale varies between 39 and 115. A high score on the scale means that the person's quality of life is high.
Quality of Life Assessment | The change scores of the patients' control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  At the end of multi-family psychoeducation, the change in the quality of life of families will be measured. Changes in health-related quality of life will be assessed with WHOQOL-BREF-TR. The scale measuring the quality of life in individuals consists of 27 items. The scale is in a 5-point Likert type and the score that can be obtained from the scale varies between 39 and 115. A high score on the scale means that the person's quality of life is high.
Depression for Families | The change scores of the families' control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  Change from baseline in Beck Depression Rating Scale at 8 weeks for families. Beck Depression Scale measuring depression in people consists of 21 items. The scale is in a 4-point Likert type and the score that can be obtained from the scale varies between 0 and 63. As the score obtained from the scale increases, the severity of depression also increases.
Depression for Patients | The change scores of the patients' control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  Change from baseline in Beck Depression Rating Scale at 8 weeks for patients. Beck Depression Scale measuring depression in people consists of 21 items. The scale is in a 4-point Likert type and the score that can be obtained from the scale varies between 0 and 63. As the score obtained from the scale increases, the severity of depression also increases.
Anxiety for Patients | The change scores of the patients' control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  Change from baseline in Beck Anxiety Rating Scale at 8 weeks for patients. Beck Anxiety Scale measuring anxiety in individuals consists of 21 items. The scale is in a 4-point Likert type and the score that can be obtained from the scale varies between 0 and 63. As the score obtained from the scale increases, the severity of anxiety also increases.
Anxiety for Families | The change scores of the families' control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  Change from baseline in Beck Anxiety Rating Scale at 8 weeks for families. Beck Anxiety Scale measuring anxiety in individuals consists of 21 items. The scale is in a 4-point Likert type and the score that can be obtained from the scale varies between 0 and 63. As the score obtained from the scale increases, the severity of anxiety also increases.
Stress Coping Skills | The change scores of the control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  The ways families cope with stress will be measured by The Ways of Coping Questionnaire.
  The scale, which measures the ways of coping with stress in individuals, consists of 30 items. The scale is in a 4-point Likert type and the score that can be obtained from the scale varies between 30 and 120. A high score on the scale means that the person is unsuccessful in terms of coping with stress.
Self Stigma for Families | The change scores of the control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  The self-stigma of families will be measured with the Self-Stigma Inventory for Families of Patients with Schizophrenia (SSI-F). There is no culturally sensitive self-stigmatization scale developed in Turkish for substance-related disorders. It is thought that this scale, which was developed for the families of schizophrenia patients, can also be used for substance-related disorders.
  The scale, which measures self-stigmatization or internalized stigmatization in individuals with mental illness, consists of 14 items. The scale is in the 5-point liker type and as the scores obtained from the scale increase, the self-stigma of the relatives of the patient increases.
Self Stigma for Patients | The change scores of the control and intervention groups between the baseline measure and pscyhoeducation completion (estimated to be 12 weeks) will be compared.
  The patients' self-stigma will be measured with the Self-Stigma Inventory for Patients with Schizophrenia (SSI-P). There is no culturally sensitive self-stigmatization scale developed in Turkish for substance-related disorders. It is thought that this scale, which was developed for schizophrenia patients, can also be used for substance-related disorders.
  The scale, which measures self-stigmatization in individuals with mental illness, consists of 17 items. The scale is in 5-point Likert type and the scores obtained from the scale vary between 17-85. As the scores obtained from the scale increase, the self-stigmatization of the patient's relatives increases.
Group Attendance | In intervention (weeks 1 to 8)
  Multifamily group attendance for psychoeducation was calculated by summing the number of treatment sessions attended. Therefore, numbers range from 0 to 8.

CONTACTS AND LOCATIONS:
Overall Officials: Zeki Yüncü, Study Director — Ege University
Locations (1):
- Maltepe University Faculty of Medicine Hospital, Alcohol and Substance Addiction Treatment Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Copello AG, Velleman RD, Templeton LJ. Family interventions in the treatment of alcohol and drug problems. Drug Alcohol Rev. 2005 Jul;24(4):369-85. doi: 10.1080/09595230500302356. PMID 16234133
- [Background] Fiorillo A, Del Vecchio V, Luciano M, Sampogna G, De Rosa C, Malangone C, Volpe U, Bardicchia F, Ciampini G, Crocamo C, Iapichino S, Lampis D, Moroni A, Orlandi E, Piselli M, Pompili E, Veltro F, Carra G, Maj M. Efficacy of psychoeducational family intervention for bipolar I disorder: A controlled, multicentric, real-world study. J Affect Disord. 2015 Feb 1;172:291-9. doi: 10.1016/j.jad.2014.10.021. Epub 2014 Oct 22. PMID 25451428
- [Background] Lucksted A, McFarlane W, Downing D, Dixon L. Recent developments in family psychoeducation as an evidence-based practice. J Marital Fam Ther. 2012 Jan;38(1):101-21. doi: 10.1111/j.1752-0606.2011.00256.x. Epub 2011 Oct 12. PMID 22283383
- [Background] McGovern R, Smart D, Alderson H, Araujo-Soares V, Brown J, Buykx P, Evans V, Fleming K, Hickman M, Macleod J, Meier P, Kaner E. Psychosocial Interventions to Improve Psychological, Social and Physical Wellbeing in Family Members Affected by an Adult Relative's Substance Use: A Systematic Search and Review of the Evidence. Int J Environ Res Public Health. 2021 Feb 12;18(4):1793. doi: 10.3390/ijerph18041793. PMID 33673199
- [Background] McFarlane WR, Link B, Dushay R, Marchal J, Crilly J. Psychoeducational multiple family groups: four-year relapse outcome in schizophrenia. Fam Process. 1995 Jun;34(2):127-44. doi: 10.1111/j.1545-5300.1995.00127.x. PMID 7589414
- [Background] Dixon L, McFarlane WR, Lefley H, Lucksted A, Cohen M, Falloon I, Mueser K, Miklowitz D, Solomon P, Sondheimer D. Evidence-based practices for services to families of people with psychiatric disabilities. Psychiatr Serv. 2001 Jul;52(7):903-10. doi: 10.1176/appi.ps.52.7.903. PMID 11433107
- [Background] Center for Substance Abuse Treatment. Substance Abuse Treatment and Family Therapy. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2004. Report No.: (SMA) 04-3957. Available from http://www.ncbi.nlm.nih.gov/books/NBK64265/ PMID 22514845
- See also: Center for Substance Abuse Treatment. Counselor's Family Education Manual: Matrix Intensive Outpatient Treatment for People With Stimulant Use Disorders. HHS Publication No. (SMA — https://store.samhsa.gov/sites/default/files/d7/priv/sma13-4153.pdf
- See also: O'Grady, C. P., Skinner, W. J.W. (2007). A Family Guide to Concurrent Disorders. Toronto: Centre for Addiction and Mental Health — https://www.camh.ca/-/media/files/guides-and-publications/partnering-with-families-guide.pdf
- See also: Substance Abuse and Mental Health Services Administration. (2022). Supporting A Loved One Dealing Wıth Mental and/or Substance Use Disorders: Starting the Conversation. — https://www.samhsa.gov/sites/default/files/starting-the-conversation-guide.pdf